CLINICAL TRIAL: NCT03892551
Title: Triage - Symptoms and Other Predictors in an All-comer Emergency Department Population (EMERGE IV)
Brief Title: Triage - Symptoms and Other Predictors in an All-comer Emergency Department Population; (EKBB 236/13)
Acronym: EMERGE IV
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: PB_2019_00008; me19Bingisser
Record Dates: First submitted 2019-03-20; First posted 2019-03-27 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Triage Risk Stratification
Keywords: risk prediction; Electronic triage systems (ETS); undertriage; overtriage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients admitted to emergency ward: all patients admitted to the emergency ward and awaiting triage are observed
  Interventions: Other: Assessment of symptoms patients presenting when admitted to ED; Other: Reason for patient presentation at ED; Other: physicians rating of severity of illness; Diagnostic Test: Assessment of vital signs; Other: Clinical Frailty Scale; Other: Impaired mobility on presentation (IMOP); Other: Assessment of suspected diagnosis and differential diagnoses

INTERVENTIONS:
Other: Assessment of symptoms patients presenting when admitted to ED — Questionnaire with a predefined list of 35 symptoms
Other: Reason for patient presentation at ED — Exploratory interview assessing reason for patient presentation at ED
Other: physicians rating of severity of illness — numeric scale ranging from 0 (perfect condition) to 10 (extremely ill)
Diagnostic Test: Assessment of vital signs — Assessment of vital signs (heart rate, blood pressure, body temperature, respiration rate, peripheral capillary haemoglobin oxygen saturation)
Other: Clinical Frailty Scale — Assessment of frailty by Clinical Frailty Scale (CFS): assess patients' frailty level from 1, very fit, to 9, terminally ill
Other: Impaired mobility on presentation (IMOP) — Assessment of IMOP: defined as being unable to stand unaided or walk without help
Other: Assessment of suspected diagnosis and differential diagnoses — Assessment of treating physician's suspected diagnosis and differential diagnoses. Answers will be recorded in free text form.

SUMMARY:
This study is to develop a tool capable of improved risk prediction regarding the 30-day mortality. Based on vital signs, impaired mobility on presentation (IMOP), Clinical Frailty Scale (CFS) and patients' symptomatology three risk categories (low, intermediate, high risk) will be established.

DETAILED DESCRIPTION:
Most Emergency Departments (EDs) perform an initial risk stratification of patients, called Triage. Establishing a diagnosis is key for the administration of the appropriate treatment and the following disposition decision. The earlier and the more accurate the final diagnosis is established, the shorter the time to treatment and time to disposition, and thus, the more efficient the patient flow. New ways to improve diagnosis accuracy early on in patients' ED visits are needed. Although a great number of well validated and widely used triage systems exists, to this date no gold standard in triage risk stratification has been established. Most of the existing triage systems rely on the measurement of vital signs and a list of chief complaints.

This study is to develop a tool capable of improved risk prediction regarding the 30-day mortality. Based on vital signs, impaired mobility on presentation (IMOP), Clinical Frailty Scale (CFS) and patients' symptomatology three risk categories (low, intermediate, high risk) will be established.

According to acuity patients undergo triage or directly proceed to the treatment unit. Patients awaiting triage will be approached by a member of the study personnel and will be verbally informed about the study. Afterwards, patients will be interviewed asking about their symptoms and their reason for presentation. Patients in need of immediate therapy will receive therapy before start of the interview. Following the interview, patients undergo routine triage.The physician performing initial triage will be asked to rate how ill patients appear to be using a numeric scale ranging from 0 (perfect condition) to 10 (extremely ill). Treating physician's will be asked to state their suspected diagnosis as well as differential diagnoses. Follow-up to assess 30-day and 1-year mortality rate and date of death will start one year after the end of the inclusion period.

ELIGIBILITY:
Inclusion Criteria:

* patients presenting to the ED of the University Hospital Basel and awaiting triage

Exclusion Criteria:

* unwillingness to participate
* insufficient ability to communicate with the study personnel.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the ED of the University Hospital Basel over a time-course of 9 weeks from 25.03.2019 to 27.05.2019.
Sampling Method: Probability Sample
Enrollment: 7309 (Actual)
Dates: Start 2019-03-18 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
30-day mortality | within 30 days of the day of presentation to the ED
  30-day mortality is defined as death within 30 days of the day of presentation to the ED

SECONDARY OUTCOMES:
Number of hospitalizations | day of presentation to the ED
  Hospitalization is defined as the direct admission from the ED to any hospital in-patient department with a stay of over 24 hours
Number of ICU-admissions | day of presentation to the ED
  ICU-admission is defined as any direct admission to the ICU of the University Hospital of Basel
Death rate (In-hospital mortality) | from day of presentation to the ED to day of hospital discharge (assessed within 365 days of the day of presentation to the ED)
  In-hospital mortality is defined as death occurring during presentation to the ED and hospital discharge
Number of institutionalisations | within 365 days of the day of presentation to the ED
  Institutionalisation is defined as no time spent at home during 365 days following presentation

CONTACTS AND LOCATIONS:
Overall Officials: Roland Bingisser, Prof. Dr., Principal Investigator — Department of Emergency Medicine, University Hospital Basel
Locations (1):
- Department of Emergency Medicine, University Hospital Basel, Basel, Switzerland

REFERENCES:
- [Derived] Rueegg M, Nissen SK, Brabrand M, Kaeppeli T, Dreher T, Carpenter CR, Bingisser R, Nickel CH. The clinical frailty scale predicts 1-year mortality in emergency department patients aged 65 years and older. Acad Emerg Med. 2022 May;29(5):572-580. doi: 10.1111/acem.14460. Epub 2022 Apr 23. PMID 35138670
- [Derived] Kaeppeli T, Rueegg M, Dreher-Hummel T, Brabrand M, Kabell-Nissen S, Carpenter CR, Bingisser R, Nickel CH. Validation of the Clinical Frailty Scale for Prediction of Thirty-Day Mortality in the Emergency Department. Ann Emerg Med. 2020 Sep;76(3):291-300. doi: 10.1016/j.annemergmed.2020.03.028. Epub 2020 Apr 24. PMID 32336486